# COVID-19 and FFP3 Mask Study Participant Information Sheet

#### **Study title:**

How Has The Increased Need For Use of FFP3 Style Respirators During the COVID-19 Pandemic Affected Hospital Doctor's Facial Hair? Implications for Staff Safety and Welfare

#### **Invitation and brief summary**

We are writing to all current hospital doctors at Royal Cornwall Hospital to kindly take part in our research study. We are examining the effects of personal protective equipment (PPE) guidance, particularly regarding FFP3 masks, on the facial hair styles of hospital doctors during the COVID-19 pandemic.

## What's involved?

We invite you to complete an online questionnaire which takes approximately 4 minutes to complete. This will be a link in your email which will take you to a Survey Monkey Questionnaire. All responses are anonymous.

## Purpose and Background to Research

The importance of effective personal protective equipment (PPE) has been highlighted during the COVID-19 global pandemic. Part of this equipment has been the use of filtering facepieces class 3 (FFP3) masks. However, these masks require staff to be either clean shaven, or significantly shave their facial hair. In addition to this, these masks do not work on all staff, regardless of facial hair style, particularly women.

The research question is to assess whether the Public Health England guidelines for facial hair styles are being followed during this global pandemic, and if not, explore the reasons this may be the case. We expect that this has implications for staff health and wellbeing, in addition to the religious and cultural reasons for maintaining particular facial hair styles. The shortage of PPE has been nationwide, and alternative PPE exist such as hoods and we will be exploring whether this has been provided.

We want this study to be as inclusive as possible, so we are inviting all RCHT doctors of all grades, genders and facial-hair growing abilities to take part.

# What would taking part involve?

Taking part would involve completing a short questionnaire, asking you some demographic questions, questions about your PPE and fit testing status. If you grow facial hair, you will be redirected to questions asking you to pick the style which closely resembles your style, and questions asking if there are any factors affecting your facial hair, in addition to if changing your facial hair style has had an effect on your mental health or wellbeing. The questionnaire uses a logic gate, so you will not necessarily answer all of the questions on the survey if they are not applicable to you. All answers are anonymous.

## What are the possible benefits of taking part?

There are no possible benefits of taking part, but it may highlight PPE shortfalls or other results which we might be able to affect positive change for our staff.

## What are the possible disadvantages of taking part?

There are no possible disadvantages to taking part.

For further information or any questions please contact <a href="mailto:Sanjeev.sahota@nhs.net">Sanjeev.sahota@nhs.net</a>

This study is receiving no funding
This study is being organised by Royal Cornwall Hospital doctors
Our local Research and Development team have reviewed the study protocl
IRAS ID 283609

Participant Information Sheet Version 1.0 6<sup>th</sup> May 2020

## **Authors:**

Dr Sanjeev Sahota Dr Simon Gill Dr Jennifer Ridenton Dr Helen Hegarty Dr Katherine Pope